CLINICAL TRIAL: NCT04271917
Title: Surgery With Alternative Pain Management (SWAP): Analgesic Effects of Cannabidiol for Simple Tooth Extractions in Dental Patients
Brief Title: Analgesic Effects of Cannabidiol for Simple Tooth Extractions in Dental Patients
Acronym: SWAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Karen Derefinko, PhD, Assistant Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-07123-XP
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute
Keywords: cannabidiol; CBD; acute pain; alternative pain management; simple extraction
MeSH Terms: conditions — Acute Pain | interventions — Cannabidiol; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Since TAU participants will receive tablets instead of oil like the other 3 arms, the design is not completely double-blinded; however, the study will be double-blinded between the other three arms which all receive oil in a dropper vial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment As Usual (TAU) (Active Comparator): Participants will receive a 5-day supply of acetaminophen 500mg and ibuprofen 200mg.
  Instructions for use: Take one tablet of each medication at the same time every 4-6 hours as needed for pain.
  Interventions: Drug: acetaminophen 500mg and ibuprofen 200mg combo
- Placebo (Placebo Comparator): Participants will receive a 5-day supply (15mL) of inactive placebo in a dropper vial.
  Instructions for use: Place 0.5mL of oil under tongue for 30 seconds then swallow. Use every 4-6 hours as needed for pain.
  Interventions: Drug: placebo
- CBD 17mg/mL (Experimental): Participants will receive a 5-day supply (15mL) of cannabidiol 17mg/mL.
  Instructions for use: Place 0.5mL of oil under tongue for 30 seconds then swallow. Use every 4-6 hours as needed for pain.
  Interventions: Drug: cannabidiol
- CBD 37 mg/mL (Experimental): Participants will receive a 5-day supply (15mL) of cannabidiol 37mg/mL.
  Instructions for use: Place 0.5mL of oil under tongue for 30 seconds then swallow. Use every 4-6 hours as needed for pain.
  Interventions: Drug: cannabidiol

INTERVENTIONS:
Drug: cannabidiol — Use of cannabidiol as an alternative to standard of care treatment of acute pain.
  Other Names: CBD oil
  Arms: CBD 17mg/mL; CBD 37 mg/mL
Drug: placebo — Inactive placebo oil to imitate CBD oil
  Arms: Placebo
Drug: acetaminophen 500mg and ibuprofen 200mg combo — standard of care
  Arms: Treatment As Usual (TAU)

SUMMARY:
The purpose of this study is to evaluate the analgesic effects of cannabidiol for patients who have undergone simple tooth extraction. Participants will be randomized to one of four arms: treatment-as-usual (TAU), cannabidiol 17mg/mL, cannabidiol 37mg/mL, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for an operatory appointment at University of Tennessee Health Science Center College of Dentistry Oral and Maxillofacial Surgery Department
* Operation must be a simple tooth extraction which does not result in an opioid prescription
* 18 years of age or older
* Have regular and direct access to a device that can send and receive texts and willing to accept any associated charges for 24 text messages

Exclusion Criteria:

* Contraindication to ibuprofen
* Contraindication to acetaminophen
* Contraindication to cannabidiol or hemp oil
* Contraindication to peppermint oil
* Contraindication to almond or other tree nuts
* Currently taking a form of cannabidiol and unwilling to stop use for one week post surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Worst pain following surgery using Wong Baker Faces pain scale | 1-week post-op
  Self-report of participant's worst pain after surgery
Amount of medication used | 1-week post-op
  Self-report of total amount of pain medication used from participant diary
Pain levels following surgery using Wong Baker Faces pain scale | First 72 hours post-op
  Self-reported pain recorded every 2 hours between 7am-9pm by automated SMS messaging.

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Derefinko, PhD, Principal Investigator — University of Tennessee; Ammaar H Abidi, DDS, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided